CLINICAL TRIAL: NCT06481605
Title: A Novel Adaptive Anastomotic Technique for Left-sided Colonic and Rectal Resection: a Pilot, Single-center, Prospective, Case-series Study
Brief Title: A Novel Adaptive Anastomotic Technique for Left-sided Colonic and Rectal Resection
Acronym: NOVA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Carponovum AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 3902
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Colorectal Neoplasms
Keywords: Colorectal Neoplasm; Anastomosis; Surgical device
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Pilot, single-center, interventional, prospective case-series study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C-REX (Experimental): Patients will receive the C-REX device during anastomosis construction
  Interventions: Device: C-REX

INTERVENTIONS:
Device: C-REX — The C-REX is a CE-marked class IIa device consisting of an invasive surgical part, including two anastomotic rings, intended for short-term use, and surgical instruments LapAid and RectoAid for assisting the placement of the anastomotic ring to intestine. The device is supplemented with a catheter to monitor the anastomosis.
  Other Names: C-REX RectoAid Cath device

SUMMARY:
The C-REX device is design to help colorectal anastomoses construction and reduce the risk of anastomotic leak. This study aims to collect preliminary evidence on the effectiveness of C-REX a real-word setting.

DETAILED DESCRIPTION:
Despite technological advancements, the rate of anastomotic leak after left colon and rectal resection remains high. In most cases, these complications are identified only from the clinical symptoms and the delay in the diagnosis may lead to more severe outcomes. The device C-REX, developed by CarpoNovum, may help the anastomosis construction, providing at the same time a system to monitor the anastomosis until complete healing. This may lead to reduced anastomotic leak rate and severity. This study aims to collect preliminary evidence on the effectiveness of C-REX to develop a future larger multicentric trial. The objective of the study is to provide preliminary data to determine whether the C-REX device may reduce the rate and severity of anastomotic leak after left colon and high rectal resection, providing new insights on the feasibility and effectiveness of the C-REX device in a real-word setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old, men or women.
* Planned primary resection due to colorectal neoplasia (cancer or benign polyps) of the sigmoid colon or rectum (above the peritoneal reflection) that require high anterior resection as the procedure of choice.
* Patient indicated to elective minimally invasive sigmoid or high rectal resection.

Exclusion Criteria:

* Patients with pre-existing health conditions requiring surgery, such as intestinal obstruction or perforation, local or systemic infections, peritonitis, or intestinal ischemia.
* Patients with preoperative evidence of distal metastasis.
* Patients with documented intestinal or anal stenosis or other obstructions distal to the anastomosis.
* Patients who received radiation therapy to organs in abdomen or pelvis unrelated to current colorectal condition.
* Patients indicated to defunctioning ileostomy (intention to treat).
* Any condition that, in the opinion of the investigator, may interfere with the study conduction. In particular, any condition which can cause significant alteration of colonic wall thickness such as chronic and repeated infection which may impair the use of C-REX.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-31 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Radiological anastomotic leaks | 90 days after surgery
  Assess the rate of radiologically confirmed anastomotic leak in the C-REX arm

SECONDARY OUTCOMES:
Severity of anastomotic leaks | 90 days after surgery
  Assess the severity of the anastomotic leaks, classifying the events according to the International Study Group of Rectal Cancer (ISGR) criteria in the C-REX arm
Positive leak tests | Intraoperative
  Assess the rate of intraoperative positive leak tests in the C-REX arm
Positive C-REX integrity tests | Intraoperative
  Assess the rate of intraoperative positive C-REX integrity tests in the C-REX arm
Time of anastomosis construction | Intraoperative
  Assess the median time of anastomosis construction in the C-REX arm
Anastomotic stenosis | 90 days after surgery
  Assess the rate of anastomosis stenosis, as assessed by the 90-day endoscopic evaluation in the C-REX arm
Postoperative complications | 90 days after surgery
  Assess the median Comprehensive Complication Index (CCI) in the C-REX arm
Helathcare costs | 90 days after surgery
  Evaluate the median healthcare costs (direct and indirect) in the C-REX arm
Low Anterior Resection Syndrome | 90 days after surgery
  Assess the median Low Anterior Resection Syndrome (LARS) score (ranging from 0 to 40, with 21 indicating significant symtpoms) in the C-REX arm.
Investigator's satisfaction | Intraoperative
  Evaluate the grade of investigator's satisfaction in using the C-REX device by using a simple likert scale ranging from 0 (completely unsatisfaid) to 5 (completely satisfaid).

CONTACTS AND LOCATIONS:
Overall Officials: Antonino Spinelli, MD, PhD, Principal Investigator — Humanitas Research Hospital IRCCS, Rozzano-Milan
Locations (1):
- IRCCS Humanitas Research Hospital, Rozzano, MI, Italy